CLINICAL TRIAL: NCT00298818
Title: Open Label Study of Zonisamide in the Treatment of Epilepsy in Patients With Mental Retardation / Developmental Disabilities
Brief Title: Open Label Study of Zonisamide in the Treatment of Epilepsy in Patients With Mental Retardation
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Alan Ettinger, MD / Chief of LIJ Comprehensive Epilepsy Center, North Shore Long Island Jewish Health System
Other Study IDs: 02.08.035
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Epilepsy; Mental Retardation; Developmental Disabilities
Keywords: Epilepsy; Mental Retardation; Developmental Disabilities
MeSH Terms: conditions — Epilepsy; Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the efficacy and tolerability in "real-world" clinical practice, of adjunctive zonisamide treatment in adult patients with developmental disabilities and epilepsy.

DETAILED DESCRIPTION:
While a number of randomized double-blind controlled trials have demonstrated the value of zonisamide in the treatment of seizures, such studies lend limited insight into the efficacy and tolerance of zonisamide in real-world clinical practice. Furthermore, randomized trials tend to inquire about negative effects, such as adverse reactions, while positive effects such as improvement in mood, or sense of well-being are not similarly categorized. In addition, there is little information about experience with zonisamide specifically in adult patients with mental retardation (MR) / developmental disabilities (DD). Anecdotal experience suggests that zonisamide is exceptionally well-tolerated, and is associated with an improved general sense of well-being and quality of life in non-DD patients. In patients with MR/DD, observational studies that promote awareness of such distinguishing features and other aspects of efficacy are essential for guiding decision-making when prescribing antiepileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, at least 18 years of age
* Diagnosis of mental retardation
* Uncontrolled seizures or intolerable side effects from current AEDs
* Legal guardian is able to consent

Exclusion Criteria:

* Sulfa allergy
* Prior exposure to zonisamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Epilepsy center
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2002-08; Primary Completion 2005-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ettinger, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States